CLINICAL TRIAL: NCT00955357
Title: An Open-Label, Multicenter, Multinational Study of Lacosamide as First Add-On Anti-epileptic Drug (AED) Treatment in Subjects With Partial-Onset Seizures
Brief Title: Trial to Assess Lacosamide as the First add-on Anti-epileptic Drug Treatment in Patients With Partial-onset Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP0954; 2009-011181-28 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2009-08-06; First posted 2009-08-10 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2017-07

CONDITIONS: Partial Epilepsies
Keywords: Epilepsy Treatment; Anti-epileptic drugs; Seizures; Vimpat
MeSH Terms: conditions — Epilepsies, Partial; Seizures | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Add-on (Experimental): Lacosamide added to first adequate monotherapy (no history of Antiepileptic Drug [AED] polytherapy) and epilepsy diagnosis < or = 24 months at Screening.
  Interventions: Drug: Lacosamide
- Later Add-on (Experimental): Lacosamide added to 1 to 3 Antiepileptic Drugs (AEDs) (with tentatives of at least 2 prior AED treatment regimens) and epilepsy diagnosis > or = 5 years at Screening.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Oral Lacosamide:
  Subjects Titration Phase (6 Weeks):
  Week 1 - 50 mg tablet Twice daily (bid); Week 2 - 100 mg tablet bid; Week 3 - 150 mg tablet bid; Week 4 - 200 mg tablet bid; Week 5 - 200 mg tablet bid; Week 6 - 150 mg tablet bid OR Week 6 - 200 mg tablet bid
  Maintenance Phase (24 Weeks):
  200 mg tablet bid OR 150 mg tablet bid
  Taper Phase (1 - 3 Weeks):
  50 mg tablet bid for 1 week OR 100 mg tablet bid for 1 week OR 150 mg tablet bid for 1 week
  Other Names: SPM927; Harkoseride; Vimpat

SUMMARY:
To evaluate the efficacy and safety of oral Lacosamide as first add on treatment in subjects with uncontrolled partial-onset seizures after prior treatment with a monotherapy Antiepileptic Drug (AED) regimen compared to subjects who have received treatment with at least 2 AEDs.

DETAILED DESCRIPTION:
The study consisted of 3 Periods: Period 1: a 1-week Screening Phase, Period 2: a 30-week Treatment Phase (consisting of a 6-week Titration Phase and a 24-week Maintenance Phase), and Period 3: a 3-week Taper/Safety Follow-Up Phase.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Subject has a diagnosis of epilepsy with simple partial seizures (motor component) and/or complex partial seizures with or without secondary generalization
* Currently taking adequate monotherapy (defined as a single Antiepileptic Drug (AED) for at least 28 days prior to Screening) and has no history of AED polytherapy. Prior use of rescue medication (short-term intermittent use) is acceptable
* Epilepsy diagnosis should be ≤24 months at the time of the Screening Visit
* The minimum allowed seizure frequency at any time during the 12 weeks prior to the Screening Visit is ≥3 partial-onset seizures

Group 2:

* Subject has a diagnosis of epilepsy with simple partial seizures (motor component) and/or complex partial seizures with or without secondary generalization
* Currently taking 1 to 3 AEDs, and has tried at least 2 prior AED treatment regimens (concurrently or sequentially)
* Epilepsy diagnosis should be ≥5 years at the time of the Screening Visit
* The minimum allowed seizure frequency during the 12 weeks prior to the Screening Visit is ≥1 partial-onset seizure per 28 days

Exclusion Criteria:

* Previous use of Lacosamide
* History of seizure disorder characterized primarily by isolated auras
* History of primary generalized seizures
* History of status epilepticus within last 12-months
* History of cluster seizures during the 12 week period prior to Visit 1
* Nonepileptic events, including pseudoseizures that could be confused with seizure
* Lifetime history of suicide attempt or suicidal ideation in the past 6 months
* Hypersensitivity to any component of Lacosamide
* History of drug or alcohol abuse
* History of an acute or subacutely progressive Central Nervous System (CNS) disease
* Undergone cranial surgery within the last year prior to study entry
* Concomitant treatment of Felbamate or previous Felbamate therapy within the last 6 months
* Prior or concomitant Vigabatrin use

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (109):
- United States (40):
  - 103, Irvine, California
  - 123, Rancho Mirage, California
  - 156, Clearwater, Florida
  - 157, Destin, Florida
  - 140, Hollywood, Florida
  - 161, Ocala, Florida
  - 108, Atlanta, Georgia
  - 112, Atlanta, Georgia
  - 124, Augusta, Georgia
  - 115, Macon, Georgia
  - 118, Rome, Georgia
  - 128, Flossmoor, Illinois
  - 130, Des Moines, Iowa
  - 102, Bowling Green, Kentucky
  - 117, Paducah, Kentucky
  - 107, Houma, Louisiana
  - 145, Ruston, Louisiana
  - 101, Annapolis, Maryland
  - 162, Waldorf, Maryland
  - 153, Boston, Massachusetts
  - 136, Pittsfield, Massachusetts
  - 144, Springfield, Massachusetts
  - 151, Kansas City, Missouri
  - 114, Paterson, New Jersey
  - 109, Brooklyn, New York
  - 133, Brooklyn, New York
  - 127, West Seneca, New York
  - 158, Charlotte, North Carolina
  - 139, Bismarck, North Dakota
  - 134, Akron, Ohio
  - 150, Canton, Ohio
  - 141, Tulsa, Oklahoma
  - 121, Indiana, Pennsylvania
  - 120, Columbia, South Carolina
  - 149, Orangeburg, South Carolina
  - 152, Spartanburg, South Carolina
  - 148, Austin, Texas
  - 154, Dallas, Texas
  - 146, Tomball, Texas
  - 119, Fredericksburg, Virginia
- 503, Vienna, Austria
- Bulgaria (9):
  - 703, Blagoevrad
  - 706, Pleven
  - 700, Sofia
  - 702, Sofia
  - 704, Sofia
  - 705, Sofia
  - 707, Sofia
  - 708, Sofia
  - 701, Varna
- Czechia (6):
  - 736, Hradec Králové
  - 735, Litoměřice
  - 733, Ostrava
  - 732, Ostrava-Hrabuvka
  - 737, Prague
  - 734, Trutnov
- 930, Aarhus, Denmark
- Finland (3):
  - 400, Helsinki
  - 402, Oulu
  - 401, Tampere
- France (2):
  - 610, Strasbourg
  - 611, Toulon
- Greece (2):
  - 521, Athens
  - 520, Thessaloniki
- Italy (10):
  - 552, Faenza
  - 546, Gallarate
  - 541, Napoli
  - 559, Pietra Ligure
  - 557, Prato
  - 540, Roma
  - 549, Roma
  - 542, Taranto
  - 547, Torino
  - 551, Trieste
- Mexico (12):
  - 180, Aguascalientes
  - 183, Chihuahua City
  - 185, Chihuahua City
  - 184, Ciudad Juárez
  - 189, Guadalajara
  - 181, Mexico City
  - 193, Mexico City
  - 195, Mexico City
  - 186, Monterrey
  - 187, Monterrey
  - 188, Monterrey
  - 182, Polanco
- Romania (4):
  - 815, Bucharest
  - 810, Cluj-Napoca
  - 814, Oradea
  - 813, Târgu Mureş
- Russia (4):
  - 830, Kazan'
  - 831, Kazan'
  - 834, Moscow
  - 833, Novosibirsk
- Spain (7):
  - 598, Terrassa, Barcelona
  - 592, Almería
  - 597, Bajo Sevilla
  - 590, Barcelona
  - 596, Santiago de Compostela
  - 594, Valencia
  - 599, Valladolid
- 892, Lausanne, Switzerland
- Turkey (Türkiye) (7):
  - 713, Adana
  - 714, Ankara
  - 710, Eskişehir
  - 711, Istanbul
  - 719, Istanbul
  - 717, Izmir
  - 718, Trabzon

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An estimated 656 subjects were to be enrolled in the study at approximately 130 sites in the US, Europe, and the rest of the world.
Pre-assignment Details: Overall 461 subjects were enrolled. The Participant Flow refers to the Safety Set (SS) which was defined as all enrolled subjects who took at least 1 dose of Lacosamide. Reasons for discontinuation were only calculated for the SS. 456 subjects were included in the Safety Set.
Groups:
- First Add-on: Lacosamide added to first adequate monotherapy (no history of Anti-Epileptic Drug [AED] polytherapy) and epilepsy diagnosis < or = 24 months at Screening.
  Lacosamide: oral tablet
  Subjects Titration Phase (6 Weeks): Week 1 - 50 mg tablet twice daily (bid); Week 2 - 100 mg tablet bid; Week 3 - 150 mg tablet bid; Week 4 - 200 mg tablet bid; Week 5 - 200 mg tablet bid; Week 6 - 150 mg tablet bid OR Week 6 - 200 mg tablet bid
  Maintenance Phase (24 Weeks): 200 mg tablet bid OR 150 mg tablet bid
  Taper Phase (1 - 3 Weeks): 50 mg tablet bid for 1 week OR 100 mg tablet bid for 1 week OR 150 mg tablet bid for 1 week
- Later Add-on: Lacosamide added to 1 to 3 Anti-Epileptic Drugs (AEDs) (with tentatives of at least 2 prior AED treatment regimens) and epilepsy diagnosis > or = 5 years at Screening.
  Lacosamide: oral tablet
  Subjects Titration Phase (6 Weeks): Week 1 - 50 mg tablet twice daily (bid); Week 2 - 100 mg tablet bid; Week 3 - 150 mg tablet bid; Week 4 - 200 mg tablet bid; Week 5 - 200 mg tablet bid; Week 6 - 150 mg tablet bid OR Week 6 - 200 mg tablet bid
  Maintenance Phase (24 Weeks): 200 mg tablet bid OR 150 mg tablet bid
  Taper Phase (1 - 3 Weeks): 50 mg tablet bid for 1 week OR 100 mg tablet bid for 1 week OR 150 mg tablet bid for 1 week
Period: Titration Phase
Arm/Group | First Add-on | Later Add-on
Started | 96 | 360
Completed | 80 | 294
Not Completed | 16 | 66
Not completed — Adverse Event | 9 | 46
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 3 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Prohibited Antiepileptic Drug change | 0 | 1
Not completed — Study medication not tolerated | 0 | 1
Not completed — Non compliance to study procedures | 0 | 1
Period: Maintenance Phase
Arm/Group | First Add-on | Later Add-on
Started | 80 | 294
Completed | 68 | 249
Not Completed | 12 | 45
Not completed — Adverse Event | 3 | 23
Not completed — Lack of Efficacy | 0 | 4
Not completed — Protocol Violation | 2 | 6
Not completed — Lost to Follow-up | 2 | 7
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Patient moving out of area | 0 | 1
Not completed — Non compliance to study procedures | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Safety Set (SS) which includes all enrolled subjects who took at least one dose of study medication. 5 subjects at one site were excluded from the Safety Set due to significant study conduct deficiencies.
Groups:
- First Add-on: Lacosamide added to first adequate monotherapy (no history of AED polytherapy) and epilepsy diagnosis < or = 24 months at Screening.
  Lacosamide: oral tablet
  Subjects Titration Phase (6 Weeks): Week 1 - 50 mg tablet twice daily (bid); Week 2 - 100 mg tablet bid; Week 3 - 150 mg tablet bid; Week 4 - 200 mg tablet bid; Week 5 - 200 mg tablet bid; Week 6 - 150 mg tablet bid OR Week 6 - 200 mg tablet bid
  Maintenance Phase (24 Weeks): 200 mg tablet bid OR 150 mg tablet bid
  Taper Phase (1 - 3 Weeks): 50 mg tablet bid for 1 week OR 100 mg tablet bid for 1 week OR 150 mg tablet bid for 1 week
- Later-Add-on: Lacosamide added to 1 to 3 AEDs (with tentatives of at least 2 prior AED treatment regimens) and epilepsy diagnosis > or = 5 years at Screening.
  Lacosamide: oral tablet
  Subjects Titration Phase (6 Weeks): Week 1 - 50 mg tablet twice daily (bid); Week 2 - 100 mg tablet bid; Week 3 - 150 mg tablet bid; Week 4 - 200 mg tablet bid; Week 5 - 200 mg tablet bid; Week 6 - 150 mg tablet bid OR Week 6 - 200 mg tablet bid
  Maintenance Phase (24 Weeks): 200 mg tablet bid OR 150 mg tablet bid
  Taper Phase (1 - 3 Weeks): 50 mg tablet bid for 1 week OR 100 mg tablet bid for 1 week OR 150 mg tablet bid for 1 week
- Total: Total of all reporting groups
Arm/Group | First Add-on | Later-Add-on | Total
Number analyzed (Participants) | 96 | 360 | 456
Age, Continuous [Median (Full Range); unit: years] | 37.5 [18.0 to 82.0] | 38.0 [16.0 to 74.0] | 38.0 [16.0 to 82.0]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 7 | 11
  Between 18 and 65 years | 82 | 349 | 431
  >=65 years | 10 | 4 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 180 | 233
  Male | 43 | 180 | 223
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 6 | 17
  Asian | 0 | 12 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 19 | 20
  White | 79 | 278 | 357
  More than one race | 5 | 45 | 50
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 99 | 123
  Not Hispanic or Latino | 72 | 261 | 333
  Unknown or Not Reported | 0 | 0 | 0
Weight [Median (Full Range); unit: kilogram] | 71.8 [42.0 to 132.9] | 73.0 [41.9 to 147.4] | 73.0 [41.9 to 147.4]
Height [Median (Full Range); unit: centimeter] | 166.5 [149.0 to 186.0] | 167.6 [140.0 to 197.0] | 167.6 [140.0 to 197.0]
BMI [Median (Full Range); unit: kilogram per m^2] | 25.3 [14.5 to 42.5] | 25.5 [17.3 to 53.9] | 25.4 [14.5 to 53.9]

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Achieved "Seizure-free Status" During the First 12 Weeks of the Maintenance Phase
Description: A subject will be considered seizure-free if the subject completes the first 12 weeks of the Maintenance Phase, reports zero seizures, and has no seizure data missing for any day during the period of time.
  This study was intended to assess the efficacy outcomes in the First Add-On Group and the Later Add-On Group individually relative to historical data. Comparisons between the 2 groups should not be attempted and conclusions should not be drawn.
Time Frame: From Week 7 (end of Week 6) to end of Week 18
Population: The Analysis Population refers to the Completer Set (CS) which includes all subjects who were enrolled, received at least one dose of Lacosamide and completed the first 12 weeks of the Maintenance Phase.
Measure: Number; unit: percentage of subjects
Groups:
- Later Add-on: Lacosamide added to 1 to 3 AEDs (with tentatives of at least 2 prior AED treatment regimens) and epilepsy diagnosis > or = 5 years at Screening.
  Lacosamide: oral tablet
  Subjects Titration Phase (6 Weeks): Week 1 - 50 mg tablet twice daily (bid); Week 2 - 100 mg tablet bid; Week 3 - 150 mg tablet bid; Week 4 - 200 mg tablet bid; Week 5 - 200 mg tablet bid; Week 6 - 150 mg tablet bid OR Week 6 - 200 mg tablet bid
  Maintenance Phase (24 Weeks): 200 mg tablet bid OR 150 mg tablet bid
  Taper Phase (1 - 3 Weeks): 50 mg tablet bid for 1 week OR 100 mg tablet bid for 1 week OR 150 mg tablet bid for 1 week
Arm/Group | First Add-on | Later Add-on
Number analyzed (Participants) | 72 | 261
percentage of subjects | 37.5 | 14.9

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were collected from Screening (Week -1) until the end of the study ( up to Week 33).
Description: Treatment Emergent Adverse Events started on/after the date of first dose and within 30 days of the date of last dose.
Arm/Group | First Add-on | Later Add-on
Serious Adverse Events (participants affected / at risk) | 8/96 | 19/360
Other Adverse Events (participants affected / at risk) | 53/96 | 212/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Add-on (N=96) | Later Add-on (N=360)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Add-on (N=96) | Later Add-on (N=360)
Vertigo (Ear and labyrinth disorders) | 9 (11) | 22 (22)
Vision blurred (Eye disorders) | 2 (3) | 24 (28)
Diplopia (Eye disorders) | 7 (7) | 17 (17)
Nausea (Gastrointestinal disorders) | 8 (8) | 24 (27)
Influenza (Infections and infestations) | 5 (5) | 4 (4)
Dizziness (Nervous system disorders) | 30 (37) | 119 (159)
Somnolence (Nervous system disorders) | 6 (8) | 54 (65)
Headache (Nervous system disorders) | 13 (19) | 41 (57)
Tremor (Nervous system disorders) | 3 (3) | 22 (23)
Anxiety (Psychiatric disorders) | 6 (6) | 4 (4)

LIMITATIONS AND CAVEATS:
This study was intended to assess the efficacy outcomes in the First Add-On Group and the Later Add-On Group individually relative to historical data. Comparisons between the 2 groups should not be attempted and conclusions should not be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days